CLINICAL TRIAL: NCT01615315
Title: Aspirin and the Risk of Microscopic Hematuria in Asymptomatic Screened Population
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sang Eun Lee, Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-URO-2012-01
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Asymptomatic General Population; Microscopic Hematuria
Keywords: aspirin; screening; microscopic hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aspirin can increase the risk of bleeding tendency. However, correlation between aspirin treatment and hematuria in general population is not well known. The investigators will evaluate whether daily use of aspirin increase the risk of microscopic hematuria in healthy large screened populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years, male or female

Exclusion Criteria:

* No result of urinalysis
* No record of medical history (including medication)

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic general population who underwent general health screening program
Sampling Method: Non-Probability Sample
Enrollment: 60048 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of the microscopic hematuria | at the screening
  >4 RBC/HPF in urine microscopy

SECONDARY OUTCOMES:
Detection rate of significant cause for microscopic hematuria | whitin 12 months after screening
  * Among participants who had microscopic hematuria at the screening
  * By imaging study or cystoscopy
  * At the screening or within 12 months after screening
  * Significant cause for microscopic hematuria
    1. urinary stone
    2. renal mass (benign or malignant / not simple cyst)
    3. urothelial cancer
    4. other lesions (clinically relevant lesions determined by researchers)
Incidence rate of persistent microscopic hematuria | within 12 months
  * Among participants who had microscopic hematuria at the screening
  * Determined by repeated urine microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sang Eun Lee, selee@snubh.org, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea